CLINICAL TRIAL: NCT00858663
Title: A Phase I Study of Radiation Therapy (IMRT) + RAD001 (Everolimus) + Cisplatin for Patients With Head and Neck Cancer
Brief Title: Radiation Therapy (IMRT) + RAD001 (Everolimus) + Cisplatin for Patients With Head and Neck Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-138
Record Dates: First submitted 2009-03-06; First posted 2009-03-10 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2013-07

CONDITIONS: Head and Neck Cancer
Keywords: RAD001(Everolimus); Cisplatin; 08-138
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Radiotherapy, Intensity-Modulated; Everolimus; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemoradiation (Experimental): * IMRT, 1 fraction/day, over approximately 33 treatment days
  * RAD001 per oral or PEG, per dose escalation scheme (Days 1 - 42)
  * Cisplatin IV weekly, per dose escalation scheme (Days 1, 8, 15, 22, 29, 36)
  Interventions: Radiation: intensity modulated radiation therapy; Drug: RAD001 (everolimus) + Cisplatin

INTERVENTIONS:
Radiation: intensity modulated radiation therapy — All patients will receive standard treatment with definitive radiation therapy (IMRT, intensity modulated radiation therapy), administered as one fraction per day (Monday through Friday) over approximately 33 fractions. Patients with resected tumors will be treated to a maximum dose of 66 Gy. Patients with unresected tumors will be treated to a maximum dose of 70 Gy.
  Patients will receive daily RAD0001 it will be administered orally or via percutaneous gastrostomy tube (PEG) once daily according to the dose escalation scheme plus cisplatin intravenously once per week (Days 1, 8, 15, 22, 29, 36) according to the dose escalation scheme.
  Approximately 3 - 4 months after completion of chemoradiation, radiologic response assessment will be performed. This will include cross-sectional imaging of the primary tumor (with CT scan and/or MRI) as well as a whole body FDG-PET (fluorodeoxyglucose positron emission tomography) scan.
Drug: RAD001 (everolimus) + Cisplatin — All patients will receive standard treatment with definitive radiation therapy (IMRT, intensity modulated radiation therapy), administered as one fraction per day (Monday through Friday) over approximately 33 fractions. Patients with resected tumors will be treated to a maximum dose of 66 Gy. Patients with unresected tumors will be treated to a maximum dose of 70 Gy.
  Patients will receive daily RAD0001 it will be administered orally or via percutaneous gastrostomy tube (PEG) once daily according to the dose escalation scheme plus cisplatin intravenously once per week (Days 1, 8, 15, 22, 29, 36) according to the dose escalation scheme.
  Approximately 3 - 4 months after completion of chemoradiation, radiologic response assessment will be performed. This will include cross-sectional imaging of the primary tumor (with CT scan and/or MRI) as well as a whole body FDG-PET (fluorodeoxyglucose positron emission tomography) scan.

SUMMARY:
The purpose of this study is to determine the best doses of RAD001 (everolimus) tablets and cisplatin to give to patients who are receiving radiation therapy for head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed head and neck carcinoma, any histology (other than sarcoma, lymphoma, or melanoma). Patients with thyroid cancer (papillary, follicular, undifferentiated, Hurthle cell, medullary, or anaplastic) may be eligible.
* Patients with cutaneous squamous cell cancer or basal cell cancer arising in the head and neck may be eligible.
* Patients will have either Stage III- IVB unresected disease (Patients with stage II-IV B hypopharynx cancer and patients with Stage IIB - IVB nasopharynx cancer may also be eligible) OR
* Will be status post macroscopically complete resection of disease with one of the following poor risk features in the surgical pathology specimen:

Malignant involvement of 2 or more regional lymph nodes Extracapsular extension of nodal disease Microscopically involved mucosal margins of resection T3 or T4 pathologic stage (excluding T3N0 laryngeal squamous cell cancer) Perineural involvement Oral cavity or oropharyngeal primaries with nodal disease at levels IV or V

* Age > or = to 18 years
* Karnofsky performance status > or = to 70%
* Adequate bone marrow function: Absolute neutrophil count > than or = to 1.5 X 109/L, Platelets > or = to 100 x 109/L, Hemoglobin > 10 g/dL.
* Adequate liver function: serum bilirubin < or = to 1.5 X upper limit of normal(ULN), and serum transaminases (alanine aminotransferase, ALT; aspartate aminotransferase, AST) activity < or = to 2.0 X ULN.
* Adequate renal function: serum creatinine within institutional normal limits, or calculated creatinine clearance (by Cockcroft and Gault method) > or = to 45 mL/min for patients with creatinine limits above institutional normal.
* INR < 1.5 or aPTT < 1.5 X upper limits of normal
* For women of child-bearing potential, negative urine or serum pregnancy test within 14 days prior to administration of RAD001.
* Men and women of childbearing potential must be willing to consent to using effective birth control methods while on treatment and for at least 3 months there after.
* The planned radiation therapy treatment dose must meet protocol requirements (Resected tumors/post-operative patients: maximum planned dose 66 Gy. Unresected tumors: maximum planned dose 70 Gy).

Exclusion Criteria:

* Any prior radiation therapy for head and neck cancer. Any prior radiation therapy to >25% of the bone marrow. Any prior radiation to whole pelvis and/or brain.
* Patients with unresected squamous cell cancer (SCC) arising in the oral cavity, oropharynx, larynx, or hypopharynx are excluded, unless they at have received at least 2 cycles of induction chemotherapy with a regimen that includes cisplatin or carboplatin. (For patients with unresected head and neck tumors other than SCC of oral cavity, oropharynx, larynx, or hypopharynx, there is no requirement for induction chemotherapy prior to protocol chemoradiation)..
* Therapeutic anticoagulation with coumadin (warfarin)
* Peripheral neuropathy > or = to grade 3, according to Common Terminology Criteria for Adverse Events (CTCAE), version 3.0.
* Hypertriglyceridemia > or = to grade 2 (CTCAE version 3.0).
* Patients who require chronic treatment with steroids ( > prednisone 5 mg/day) or other immunosuppressive agents are excluded. Both cisplatin and RAD001 are immunosuppressive, and chronic steroid use (> prednisone 5 mg/day) or use of other immunosuppressive agents might increase the risk of lethal infection in this setting. Patients on low- dose steroid replacement regimens (< or = to prednisone 5 mg/day) are not excluded, because low dose steroids should not be immunosuppressive.
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001 (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection).
* Active infection or serious underlying medical condition that would impair the patient's ability to receive protocol treatment. Other concurrent severe and/or uncontrolled medical disease which would compromise participation in the study in the opinion of the investigator (e.g., uncontrolled diabetes, unstable angina, or congestive heart failure - New York Heart Association Class III or IV)
* HIV-positive patients. These patients are at increased risk of lethal infections when treated with marrow suppressive therapy. Additionally, pharmacokinetic interactions between antiretroviral therapy and the study regimen may be problematic for these patients.
* Women who are pregnant or lactating
* Other active malignancy, other than indolent malignancies which the investigator determines are unlikely to interfere with treatment and safety analysis. For example, patients with nonmelanoma skin cancer, in situ carcinoma of the cervix, or prostate cancer with no current biochemical (PSA) or radiologic evidence of disease may enroll.
* Impaired lung function: O2 saturation 88% or less at rest on room air by Pulse Oximetry. If O2 saturation is < or = to 88% at rest, further pulmonary function tests (PFTs) should be ordered to confirm normal pulmonary function and eligibility.
* Patients should not receive immunization with attenuated live vaccines within one week of study entry or during the study period. Close contact with those who have received attenuated live vaccines should be avoided during treatment with everolimus. Examples of live vaccines include intranasal influenza, measles, mumps, rubella, oral polio, BCG, yellow fever, varicella, and TY21a typhoid vaccines.
* Liver disease such as cirrhosis or severe hepatic impairment (Childs-Pugh class C).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-03; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
To establish the phase II recommended dose of oral RAD001 (everolimus) tablets + weekly intravenous cisplatin given concurrently with radiation therapy. | 3 months

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of oral RAD001 + radiation therapy + intravenous cisplatin. | 3 months
To estimate the incidence of over-expression of eIF4E in surgical margins by immunohistochemistry (IHC).(only for those subjects who undergo primary surgery) | 3 months
To describe the pharmacokinetics of RAD001 administered by PEG (percutaneous gastrostomy) tube. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Fury, MD,PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org